CLINICAL TRIAL: NCT02653274
Title: Gastrointestinal and Blood Glucose Responses to Breakfast Porridges Made From Different Grains: A Magnetic Resonance Imaging Pilot Study in Healthy Volunteers
Brief Title: Assessment of Millet, Oat and Rye Porridge Breakfasts Glucose and Gastric Emptying
Acronym: AMORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: F14072015 SoM SPMIC BMedSci
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: MRI; blood glucose; satiety; breakfast; porridge; grains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- OATS PORRIDGE (Active Comparator): Oats breakfast porridge
  Interventions: Other: Breakfast porridge
- RYE PORRIDGE (Active Comparator): Rye breakfast porridge
  Interventions: Other: Breakfast porridge
- FINGER (RAGI) MILLET PORRIDGE (Active Comparator): Finger (ragi) millet breakfast porridge
  Interventions: Other: Breakfast porridge
- PEARL (BAJRA) MILLET PORRIDGE (Active Comparator): Pearl (bajra) millet breakfast porridge
  Interventions: Other: Breakfast porridge

INTERVENTIONS:
Other: Breakfast porridge — 220 kcal breakfast porridge served with 240 mL glass of water

SUMMARY:
Breakfast porridges are made from milled grains and are commonly eaten worldwide. Traditionally different grains are used in different countries. For example, oats are more common in the Anglo-Saxon countries; rye is favoured in the Scandinavian countries whilst millet is very common in parts of India and Africa. However the nutritional value and potential metabolic and health effects may vary dramatically between different grains. For example what is the effect of the different grains on blood sugar or on how fast the stomach empties after eating the porridge and how full people feel. All these physiological responses may differ between these grains resulting in potential health benefits.

RESEARCH QUESTION: The investigators hypothesise that porridges made from different grains will behave differently during the digestion and cause differences in blood glucose levels, gastric emptying and appetite.

This study, which is a 4-way, randomized, cross over pilot study in healthy participants, aims to answer this research question.

The participants will be asked to eat a porridge breakfasts made with oats, rye and millet of different varieties (but containing the same amount of calories), in 4 morning studies one week apart. MRI will be used to monitor the gastrointestinal fate of the breakfasts and measure gastric emptying using MRI, blood glucose levels using a finger prick test and self-reported appetite scores.

DETAILED DESCRIPTION:
Background: Porridge breakfasts from various grains are a staple source of energy for many populations worldwide. The grains used in the porridges differ between regions, mostly due to the crops historically grown. For example, oats are more common in the Anglo-Saxon countries; rye is traditional in the Scandinavian countries whilst millet is very common in parts of India and Africa. Porridge consumption is very popular: 78% of South Africans eat porridge; 49% of British people eat porridge with 23% doing so almost daily; 62% of U.S. households buy hot cereal breakfast and the hot cereal segment is the best performer within the breakfast cereals market in the UK. Consumption of whole grains has been associated with a variety of health benefits ranging from lower blood glucose levels, improved insulin responses, reduced cholesterol and increased diversity of the microbiota. Of particular interest to this study are recent suggestions that different grains, and particularly millet grains, may have enhanced health benefits on glucose and insulin metabolism. This may be due to different rates of digestion and absorption, for example, because of grain specific differences in starch digestibility. This could affect gastric emptying and, in turn, post prandial glycaemia and impact on satiety. However little is known about possible differences in gastric emptying between breakfast porridges from different grains and possible relationship with glucose, insulin and appetite.

The hypothesis underlying this study is that porridges made from different grains (such as oats, rye and different millets) will produce different postprandial glucose levels and that these will correlate with gastric emptying and appetite in healthy volunteer participants.

Aims: 1. to collect pilot data on postprandial glucose levels of isoenergetic breakfast porridges made from different grains, such as oats, rye and millets of different origin. 2. to collect initial pilot data on their gastric emptying and satiety. 3. to compare postprandial glucose levels, gastric emptying and satiety for the different treatments 4. to explore relationships between glucose levels, gastric emptying and satiety.

Experimental protocol and methods: 16 healthy volunteers will participate in this 4-way study. They will attend one morning for each study, with the studies separated by 1 week. Before the test meal, and after that approximately every 15 min for 1 hour and after that approximately every 20 minutes for 1 hour the level of glucose in their blood will be measured using the finger prick method, as diabetics commonly do to monitor their blood sugars. The participants will also be scanned at baseline, immediately after the test meal and then every hour for 2 hours postprandially. Subjects will be scanned on a research dedicated 1.5T MRI scanner. At baseline and every time the subjects provide a blood glucose sample the participants will be asked to rate their feelings of fullness, hunger and appetite on 100mm VAS scales.

The subject will be fed four isoenergetic breakfast porridges: Oat, Rye, Pearl (Bajra) millet and Finger (Ragi) millet porridge sourced from supermarkets or food shops. These will be cooked in water to avoid confounding factor with milk. The test breakfast will have 220 kcal.

Statistical power. This is only a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2
* Able to give informed consent
* Apparently healthy: no medical conditions which might affect study measurements (judged by study physician)

Exclusion Criteria:

* Use of medication which interferes with study measurements (as judged by the study physician).
* Participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study.
* Not used to eating breakfast
* Not used to eating three meals a day
* Reported participation in night shift work during the two weeks prior to pre-study investigation or during the study. Night work is defined as working between midnight and 6.00 AM.
* Strenuous exercise for more than10 hours per week.
* Consumption of ≥21 alcoholic drinks in a typical week
* Reported weight loss or gain ≥ 10 % of bodyweight during the six months period before the pre-study examination.
* Following a medically- or self-prescribed diet during the two weeks prior to the pre-study examination and until the end of the study
* Dislike of the products served as the dietary test treatments
* Any allergy or food intolerance to the test treatments
* An eating disorder as indicated by the Three factor eating questionnaire
* Not suitable for MRI scanning (e.g., presence of metal implants, infusion pumps and pacemakers) as assessed by standard MRI safety questionnaire.
* Pregnancy declared by candidate
* Antibiotic or prescribed probiotic treatment in the past 12 weeks
* Inability to lie flat
* Exceeding the scanner bed weight limit of120kg
* Poor understanding of the spoken and/or written English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | From baseline up to 2 hours postprandially
  Area Under the Curve of post prandial blood glucose, measured using finger prick method, up to 2h (AUC2h) postprandially

SECONDARY OUTCOMES:
Gastric volumes | From baseline up to 2 hours postprandially
  Area Under the Curve of post prandial gastric volumes, measured by MRI, up to 2h (AUC2h) postprandially

OTHER OUTCOMES:
Time to peak of blood glucose | From baseline up to 2 hours postprandially
  Time to peak of post prandial blood glucose, measured using finger prick method, up to 2h (AUC2h) postprandially
Appetite VAS | From baseline up to 3 hours postprandially
  Area Under the Curve for appetite (Fullness, Hunger, Prospective food consumption) post prandial 100 mm VAS scores AUC2h and AUC 3h
Small bowel water content | From baseline up to 2 hours postprandially
  Area Under the Curve of post prandial small bowel water content, measured by MRI, up to 2h (AUC2h) postprandially
Food diaries | From 12:00 hours to 22:00 hours on the study day
  Records of all food eaten on the study day beyond the breakfast porridge provided in the morning
Correlations between blood, MRI and satiety data | From baseline up to 2 hours postprandially
  Exploratory correlations between blood, MRI and satiety data

CONTACTS AND LOCATIONS:
Overall Officials: Jaber Alyami, MRes, Study Director — Nottingham Digestive Diseases Centre
Locations (1):
- Nottingham Digestive Disases Centre, Nottingham, Nottinghamshire, United Kingdom